CLINICAL TRIAL: NCT02041169
Title: Lower Extremity Peripheral Arterial Disease and Exercise Ischemia: Walking Capacity Variability, Pain Evolution and Pathophysiological Responses. The CLASH Study.
Brief Title: Lower Extremity Peripheral Arterial Disease and Exercise Ischemia
Acronym: CLASH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 35RC13-9907-CLASH; 2013-A01381-44 (Other: ANSM); 13/34-914 (Other: CPP Ouest V)
Record Dates: First submitted 2014-01-14; First posted 2014-01-20 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Peripheral Arterial Diseases; Intermittent Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Subsequent walking performance (Experimental): Subsequent walking performance
  Interventions: Other: Subsequent walking performance

INTERVENTIONS:
Other: Subsequent walking performance — Subsequent walking performance

SUMMARY:
Lower extremity peripheral arterial disease (LEPAD) is a highly prevalent chronic disease. Cardiovascular mortality of LEPAD patients at five years ranges between 18 to 30%. LEPAD is primarily caused by atherosclerosis that induces an inadequate blood flow to meet the tissues demand due to the narrowing of the arteries. An aggravation of the arterial lesions in LEPAD patients induces a worsening of patients' symptoms and a severe limitation of their walking capacity, contributing to an impairment of their quality of life. Despite maintaining a sufficient walking activity is essential for these patients, LEPAD patients lower their physical activity, which worsen the disease and potentially contribute to increase the risk of cardiovascular events and deaths.

In a recent study in LEPAD patients, we showed, from a one hour GPS recording, a high variability of the patients' walking capacity (i.e., walking distances between two stops induced by lower limbs pain). Results suggested that in most patients previous stop duration before each walk was a predictor parameter of this walking variability. Whether there is an optimal or minimal recovery time influencing the walking capacity in LEPAD patients has never been studied.

This study is a prospective, cross-sectional study in exercise pathophysiology.

The main goal is to determine, following a walk that induces ischemia, the influence of the recovery duration on the subsequent walking performance in LEPAD patients.

Secondary goals are :

1. To determine the nature of the relationship between the recovery duration and subsequent walking performance.
2. To study the relationship between exercise ischemia, pain evolution and previous recovery duration.
3. To determine whether the experimental procedure influence the determination of an optimal of minimal recovery duration.
4. To study the influence of recovery duration on walking capacity from community-based measurement.

DETAILED DESCRIPTION:
It is expected to determine for the first time an optimal recovery duration that would maximize the walking capacity of LEPAD patients.

In the medium term :

* To give indications to the LEPAD patients to manage their pain in the community without lower their physical activity.
* To limit the functional decline of LEPAD patients.
* To influence the quality of life and cardiovascular mortality. This would deserve furthers studies.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Insured under the French social security system (according to French law)
* Presence of lower-extremity peripheral artery disease, defined by:

  * A resting ankle-brachial index (ABI) ≤ 0.90
  * OR if resting ABI > 0.90 and < 1.00, a decrease in recovery ankle systolic pressure or in recovery ABI from treadmill exercise higher than 30% or 20%, respectively (AHA recommendations).
  * OR if resting ABI > 1.40, a toe pressure index ≤ 0.70
* Maximal walking distance on treadmill (3.2 km/h, 10% grade) < 500m (a)
* Complain of exertional lower limbs pain that can begin or not at rest, causes the participant to stop walking and relieves or lessens within 10 minutes of rest (assessed using the San Diego questionnaire AND confirmed during treadmill testing) (b)

  1. As assessed during the medical appointment.
  2. According to our inclusion criteria, patients' leg symptoms that fell within the following leg symptom categories could be included in the study:

  i) Intermittent claudication. Patients that experience exertional calf pain that does not begin at rest and that forces them to stop walking and that relieves or lessens within 10 minutes of rest; ii) Atypical exertional leg pain/stop. This category can encompass diverse situations of exertional leg symptoms. In the present study, patients in this category were included if they experience exertional pain that does not begin at rest and that forces them to stop walking, but that do not involve only the calf(s) but also thigh(s) and/or buttock(s). Further, the exertional leg pain relieves or lessens within 10 minutes of rest; iii) Leg pain on exertion and rest. In this category, patients sometimes experience exertional leg pain at rest when they are standing still or sitting. On exertion, patients also experience a walking pain as described above. As reminded by Criqui et al., this category of patients with "pain at rest" should not be confused with patients that experience "rest pain", which usually refers to patients with such severe advanced PAD that ischemic pain is present even at rest. Patients with ischemic rest pain were not included in the study.

Non-Inclusion criteria

* Exercise limitation due to symptoms not related to an arterial insufficiency in the lower limbs (e.g., dyspnea, angina pectoris)
* Contraindication for walking (Abdominal aortic aneurysm > 4 cm)
* Myocardial infarction and no stroke in the last 3 months
* Critical limb ischemia, amputation.
* Pregnant women
* Adult subject to legal protection (guardianship or tutelage measure) and persons deprived from their liberty (according to French law).
* Patient living more than 50 km from the university hospital
* Patient unable to understand the instructions of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-09 (Actual); Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Coefficient of determination between the recovery duration and subsequent walking performance, obtained from individual regression analyses. | 32 days
  Coefficient of determination between the recovery duration and subsequent walking performance, obtained from individual regression analyses.

SECONDARY OUTCOMES:
Coefficient of determination determined from different curves fitting | 32 days
  Coefficient of determination determined from different curves fitting

OTHER OUTCOMES:
Coefficient of correlation between the level of ischemia during recovery and exercise ischemia and pain occurrence during subsequent walking | 32 days
  Coefficient of correlation between the level of ischemia during recovery and exercise ischemia and pain occurrence during subsequent walking
Coefficient of correlation between the optimal recovery duration measured on the laboratory and measures from community-based measurements. | 32 days
  Coefficient of correlation between the optimal recovery duration measured on the laboratory and measures from community-based measurements

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume MAHE, MD, Principal Investigator — Rennes University Hospital
Locations (1):
- Rennes University Hospital, Rennes, Brittany Region, France

REFERENCES:
- [Result] de Mullenheim PY, Chaudru S, Mahe G, Prioux J, Le Faucheur A. Clinical Interest of Ambulatory Assessment of Physical Activity and Walking Capacity in Peripheral Artery Disease. Scand J Med Sci Sports. 2016 Jul;26(7):716-30. doi: 10.1111/sms.12512. Epub 2015 Jul 15. PMID 26173488
- [Result] Chaudru S, Jehannin P, de Mullenheim PY, Klein H, Jaquinandi V, Mahe G, Le Faucheur A. Using wearable monitors to assess daily walking limitations induced by ischemic pain in peripheral artery disease. Scand J Med Sci Sports. 2019 Nov;29(11):1813-1826. doi: 10.1111/sms.13511. Epub 2019 Jul 31. PMID 31271680
- [Result] Donnou C, Chaudru S, Stivalet O, Paul E, Charasson M, Selli JM, Mauger C, Chapron A, Le Faucheur A, Jaquinandi V, Mahe G. How to become proficient in performance of the resting ankle-brachial index: Results of the first randomized controlled trial. Vasc Med. 2018 Apr;23(2):109-113. doi: 10.1177/1358863X17740993. Epub 2017 Nov 10. PMID 29125051
- [Result] de Mullenheim PY, Rouviere L, Emily M, Chaudru S, Kaladji A, Mahe G, Le Faucheur A. "Should I stay or should I go now?" Recovery time effect on walking capacity in symptomatic peripheral artery disease. J Appl Physiol (1985). 2021 Jul 1;131(1):207-219. doi: 10.1152/japplphysiol.00441.2020. Epub 2021 May 13. PMID 33982591